CLINICAL TRIAL: NCT03956589
Title: Functional Respiratory Imaging (FRI) to Assess the Short-term Effect of the Product ORKAMBI (Lumacaftor/ Ivacaftor) on Lung Function in ORKAMBInaive Patients With Cystic Fibrosis Homozygous for Phe508del
Brief Title: Functional Respiratory Imaging and Orkambi in CF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patient inclusion has stopped after interim analysis.
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Stijn Verhulst, Director Department of Pediatrics, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001573-24
Record Dates: First submitted 2019-05-02; First posted 2019-05-20 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orkambi open-label arm (Experimental): Open-label study: all subjects will receive Orkambi during 3 months.
  Interventions: Drug: Orkambi

INTERVENTIONS:
Drug: Orkambi — Open label of Orkambi treatment during 3 months

SUMMARY:
Open-label study to investigate the effects of Orkambi in CF patients homozygous for the F508del mutation by functional respiratory imaging. Primary endpoints in this study are the changes in Specific airway volumes (siVaw) and Specific Airway resistance (siRaw). A total of 20 ORKAMBI-naive patients with Cystic Fibrosis, homozygous for the F508del mutation will be included in this open label study and will be followed through 3 months of treatment. The treatment will be started after all assessments are performed at visit 1. After the start of the treatment some baseline measurements will be repeated throughout the 3-month treatment period. The patient will be asked to visit the hospital monthly. All study visits should be scheduled around the same time.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF (homozygous for the F508del mutation must be present, this should be documented in the medical history).
* Age ≥ 12 years
* FEV1 > 50%
* Signed informed consent. If patient is a minor, parents/guardians must give written informed consent
* Patient must be on a stable regimen of CF medication for 4 weeks prior to Visit

Exclusion Criteria:

* FEV1 < 50%
* Anticipated requirement for hospitalization within the next three weeks
* History of pneumothorax within the past 6 months prior to Visit 1
* History of haemoptysis requiring embolization within the past 12 months prior to Visit 1
* Unable or unwilling to complete study visits or provide follow-up data as required per the study protocol
* Has taken Intravenous (IV) antibiotics within the past 4 weeks prior to Visit 1
* Has ongoing exacerbation or Allergic bronchopulmonary aspergillosis (ABPA)
* Pregnant or lactating female
* Posttransplant patients
* Patients with severe hepatic impairment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in specific image-based airway resistance (siRaw) | baseline and after three months of therapy
  Change in CFD-based airway resistance normalized by the lung volume
Change in specific image-based airway volumes (siVaw) | baseline and after three months of therapy
  change in CT-based airway volumes normalized by the lung volume

SECONDARY OUTCOMES:
Internal Airflow Distribution | baseline and after three months of therapy
  calculated using thorax HRCT
Air Trapping | baseline and after three months of therapy
  calculated using thorax HRCT
Airway Wall Volume | baseline and after three months of therapy
  calculated using thorax HRCT
Aerosol Deposition | baseline and after three months of therapy
  calculated using thorax HRCT
Dynamic lung volumes | baseline and after three months of therapy
  calculated using spirometry
Static lung volumes | baseline and after three months of therapy
  calculated using body plethysmography
airway resistances | baseline and after three months of therapy
  calculated using body plethysmography
Lung clearance index | baseline and after three months of therapy
  Marker of lung ventilation inhomogeneity
6-minute walking test | baseline and after three months of therapy
  Marker of fitness for daily activities
Sweat chloride test | baseline and after three months of therapy
  Chloride values in sweat chloride test
CFQ-R | baseline and after three months of therapy
  standardized measures of quality of life will be administered to subject and to parents of subjects under 18 years of age. Disease-specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms. Developed specifically for use in patients with a diagnosis of cystic fibrosis. Scores range from 0 to 100, with higher scores indicating better health.
Digital lung auscultation | baseline and after three months of therapy
  Digital analysis of digital lung sounds obtained by a digital stethoscope
Exacerbation frequency | baseline and after three months of therapy
  Number of cystic fibrosis exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Verhulst, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No